CLINICAL TRIAL: NCT06892626
Title: Flexible Ureteroscopy Versus Percutaneous Nephrolithotomy As Primary Treatment in Renal Stones 2-3 Cm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hesham Kamal Torad, Dr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FURS-PCNL
Record Dates: First submitted 2025-03-10; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Stones, Kidney; Stones Ureter; Urolithiasis
MeSH Terms: conditions — Kidney Calculi; Ureterolithiasis; Urolithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RIRS (Experimental): RIRS performed in lithotomy position for which guide wire pass to the kidney, then passing ureteral dilators up to 14F and ureteral access sheath. Dusting stones by RIRS and holmium laser Fiber 200 mm, at the end of operation DJ was fixed.
  Interventions: Procedure: RIRS
- PNL (Experimental): PNL performed in prone position, after passing guide wire and ureteric catheter in lithotomy position. Puncture to the kidney, passing 2 wires, then using renal dilators and access sheath to enter kidney by nephroscopy, fragment stones by pneumatic and remove stones, then place nelaton 28F at end of operation.
  Interventions: Procedure: PNL

INTERVENTIONS:
Procedure: RIRS — RIRS performed in lithotomy position for which guide wire pass to the kidney, then passing ureteral dilators up to 14F and ureteral access sheath. Dusting stones by RIRS and holmium laser Fiber 200 mm, at the end of operation DJ was fixed.
  Arms: RIRS
Procedure: PNL — PNL performed in prone position, after passing guide wire and ureteric catheter in lithotomy position. Puncture to the kidney, passing 2 wires, then using renal dilators and access sheath to enter kidney by nephroscopy, fragment stones by pneumatic and remove stones, then place nelaton 28F at end of operation
  Arms: PNL

SUMMARY:
Flexible Ureteroscopy versus Percutaneous Nephrolithotomy as Primary Treatment in Renal Stones 2-3 Cm

ELIGIBILITY:
Inclusion Criteria:

stone burden from 2- 3 cm, single or multiple stones and radio-opaque or radio-lucent stones.

Exclusion Criteria:

stone burden from 2- 3 cm, single or multiple stones and radio-opaque or radio-lucent stones.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
stone free rate percentage defined as number of patients who have no stone residual | 18 months
  assessed by Plain urinary tract and ultrasound for confirmation of the presence of residual stone fragments.

CONTACTS AND LOCATIONS:
Locations (1):
- Hesham Torad, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided